CLINICAL TRIAL: NCT03265964
Title: Clinical and Imaging Biomarker Trial of Uridine for Veterans With Suicidal Ideation
Brief Title: Clinical and Imaging Trial of Uridine for Veterans With Suicidal Ideation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBB-012-16F; 00100075 (Other: Salt Lake City VAMC)
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Suicidal Ideation
Keywords: Suicidal Ideation; Veteran; Uridine; Neuroimaging
MeSH Terms: conditions — Suicidal Ideation | interventions — Uridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Uridine (Active Comparator): Subjects randomized to this study arm will receive uridine 2000 mg daily by mouth for 4 weeks
  Interventions: Drug: Uridine
- Placebo (Placebo Comparator): Subjects randomized to this arm of the study will receive placebo 2000 mg daily by mouth for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Uridine — Uridine is the active treatment in this clinical trial.
  Other Names: Oral Uridine
  Arms: Uridine
Drug: Placebo — Pill placebo is the inactive treatment comparator in this clinical trial.
  Other Names: Oral Pill Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of the investigational drug uridine as a treatment for suicidal ideation in veterans.

The investigators hypothesize that the administration of a naturally occurring dietary supplement, uridine, will rapidly reduce suicidal ideation in veterans. The purpose of this study is to determine whether 4 weeks of uridine supplementation is an effective treatment for suicidal ideation in veterans, when compared to a group taking a placebo.

DETAILED DESCRIPTION:
Veteran suicides, attempts and suicidal ideation (SI) remain an urgent concern for the Veterans Health Administration (VHA). Research indicates that approximately half of veteran suicides take place within 1 month of the decedent's final VHA encounter, with one quarter occurring within 1 week. This provides a temporal window of opportunity to intervene, and necessitates development of a rapid-acting treatment for veterans with SI. Uridine shares similar brain mechanisms and neural effects with ketamine and lithium, treatments commonly used to reduce suicidal ideation. This study will test the novel intervention uridine as a rapid-acting oral treatment for veterans with suicidal ideation. The purpose of this study is to investigate whether uridine can decrease suicidal ideation in veterans when taken daily for 4 weeks.

In addition to treatment with the investigational drug versus placebo, the study includes a translational neuroimaging component: magnetic resonance spectroscopy (1H-MRS) brain scans are performed at baseline, and then repeated following 1 week of treatment with uridine or placebo. The scans do not use radiation, and are performed on a 3 Tesla MRI system that is approved for clinical use. The scans allow researchers to measure the concentrations of several chemicals in the brain that are may be involved in suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to Provide Informed Consent.
* Must be a Veteran of the U.S. Armed Forces.
* Columbia-Suicide Severity Rating Scale Indicates Current Suicidal Ideation
* Beck Scale for Suicide Ideation Score > 3 (i.e. "Greater Than or Equal to 4").
* History of > 1 Suicide Attempt or Hospitalization to Prevent Suicide in Past 12 Months; or Functionally Impairing Suicidal Ideation Not Due to a DSM Axis II Diagnosis, in the Past 12 Months.
* Females and Males Ages 18-55 Inclusive.
* Willing and Able to Identify an Alternative Contact Person, e.g. Family Member, Friend or Neighbor.

Exclusion Criteria:

* Schizophrenia or Other Psychotic Disorder.
* Active Substance Use Disorder Requiring Stabilization (N.B. Does Not Include Nicotine).
* Unstable Medical Condition(s).
* Pregnancy or Breastfeeding.
* Contraindication to MRI (e.g. Ferrometallic Implant or Claustrophobic Anxiety).
* Concurrent Enrollment in Another Clinical Trial.
* Significant Risk of Protocol Non-Adherence (e.g. resides > 50 miles from the hospital, and has no automobile or alternate transportation).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Gavin Kondo, MD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kondo DG, Sung YH, Hellem TL, Delmastro KK, Jeong EK, Kim N, Shi X, Renshaw PF. Open-label uridine for treatment of depressed adolescents with bipolar disorder. J Child Adolesc Psychopharmacol. 2011 Apr;21(2):171-5. doi: 10.1089/cap.2010.0054. Epub 2011 Apr 12. PMID 21486171
- [Background] Agarwal N, Sung YH, Jensen JE, daCunha G, Harper D, Olson D, Renshaw PF. Short-term administration of uridine increases brain membrane phospholipid precursors in healthy adults: a 31-phosphorus magnetic resonance spectroscopy study at 4T. Bipolar Disord. 2010 Dec;12(8):825-33. doi: 10.1111/j.1399-5618.2010.00884.x. PMID 21176029
- [Background] Jensen JE, Daniels M, Haws C, Bolo NR, Lyoo IK, Yoon SJ, Cohen BM, Stoll AL, Rusche JR, Renshaw PF. Triacetyluridine (TAU) decreases depressive symptoms and increases brain pH in bipolar patients. Exp Clin Psychopharmacol. 2008 Jun;16(3):199-206. doi: 10.1037/1064-1297.16.3.199. PMID 18540779
- [Background] Carlezon WA Jr, Mague SD, Parow AM, Stoll AL, Cohen BM, Renshaw PF. Antidepressant-like effects of uridine and omega-3 fatty acids are potentiated by combined treatment in rats. Biol Psychiatry. 2005 Feb 15;57(4):343-50. doi: 10.1016/j.biopsych.2004.11.038. PMID 15705349
- [Background] Yoon SJ, Lyoo IK, Kim HJ, Kim TS, Sung YH, Kim N, Lukas SE, Renshaw PF. Neurochemical alterations in methamphetamine-dependent patients treated with cytidine-5'-diphosphate choline: a longitudinal proton magnetic resonance spectroscopy study. Neuropsychopharmacology. 2010 Apr;35(5):1165-73. doi: 10.1038/npp.2009.221. Epub 2009 Dec 30. PMID 20043005
- [Background] Wurtman RJ, Cansev M, Ulus IH. Synapse formation is enhanced by oral administration of uridine and DHA, the circulating precursors of brain phosphatides. J Nutr Health Aging. 2009 Mar;13(3):189-97. doi: 10.1007/s12603-009-0056-3. PMID 19262950
- [Background] Liu P, Wu C, Song W, Yu L, Yang X, Xiang R, Wang F, Yang J. Uridine decreases morphine-induced behavioral sensitization by decreasing dorsal striatal dopamine release possibly via agonistic effects at GABAA receptors. Eur Neuropsychopharmacol. 2014 Sep;24(9):1557-66. doi: 10.1016/j.euroneuro.2014.06.010. Epub 2014 Jun 28. PMID 25088943
- [Background] Price GD, Robertson SJ, Edwards FA. Long-term potentiation of glutamatergic synaptic transmission induced by activation of presynaptic P2Y receptors in the rat medial habenula nucleus. Eur J Neurosci. 2003 Feb;17(4):844-50. doi: 10.1046/j.1460-9568.2003.02501.x. PMID 12603274
- [Background] Wirkner K, Gunther A, Weber M, Guzman SJ, Krause T, Fuchs J, Koles L, Norenberg W, Illes P. Modulation of NMDA receptor current in layer V pyramidal neurons of the rat prefrontal cortex by P2Y receptor activation. Cereb Cortex. 2007 Mar;17(3):621-31. doi: 10.1093/cercor/bhk012. Epub 2006 Apr 28. PMID 16648456
- [Background] Saydoff JA, Garcia RA, Browne SE, Liu L, Sheng J, Brenneman D, Hu Z, Cardin S, Gonzalez A, von Borstel RW, Gregorio J, Burr H, Beal MF. Oral uridine pro-drug PN401 is neuroprotective in the R6/2 and N171-82Q mouse models of Huntington's disease. Neurobiol Dis. 2006 Dec;24(3):455-65. doi: 10.1016/j.nbd.2006.08.011. Epub 2006 Sep 29. PMID 17011205
- [Background] Tochigi M, Iwamoto K, Bundo M, Sasaki T, Kato N, Kato T. Gene expression profiling of major depression and suicide in the prefrontal cortex of postmortem brains. Neurosci Res. 2008 Feb;60(2):184-91. doi: 10.1016/j.neures.2007.10.010. Epub 2007 Nov 6. PMID 18068248
- See also: Methods of treatment of bipolar disorder [US Patent Application 20110160158 A1] — https://www.google.com/patents/US20110160158

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Uridine | Placebo
Started | 37 | 38
Completed | 32 | 35
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uridine | Placebo | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 38 | 75
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.89 (8.33) | 37.65 (7.14) | 39.29 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 31 | 30 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 34 | 31 | 65
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The hypothesis is that 4 weeks of uridine 2000 mg daily will decrease the probability and severity of suicidal ideation measured with the C-SSRS, compared with placebo. Scores range from 0 to 25 with higher scores representing more severe suicidal ideation.
Time Frame: 4 weeks
Population: Participants who were non-adherent to the study protocol or had medication changes throughout the clinical trial were removed from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Uridine | Placebo
Number analyzed (Participants) | 29 | 26
score on a scale
  Baseline: Week 0 | 13.69 (2.04) | 14.46 (2.73)
  End of Treatment: Week 4 | 8.27 (6.45) | 10.87 (5.20)

2. Primary Outcome: Change From Baseline in Beck Scale for Suicide Ideation (BSSI)
Description: The hypothesis is that 4 weeks of uridine 2000 mg daily will decrease the probability and severity of suicidal ideation measured with the BSSI compared with placebo. The BSSI is a 19 item measure on a 0-2 point scale for a range of 0-38, with higher scores indicating higher suicidal ideation or worse outcomes.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Uridine | Placebo
Number analyzed (Participants) | 29 | 26
score on a scale
  Baseline: Week 0 | 14.52 (4.26) | 17 (5.78)
  End of Treatment: Week 4 | 6.35 (6.37) | 10.57 (7.26)

3. Primary Outcome: Change From Baseline in Brain Gamma-Aminobutyric Acid (GABA)/NAA Levels, Measured With Proton-1 Magnetic Resonance Spectroscopy (1H-MRS) Neuroimaging
Description: The hypothesis is that Brain Gamma-Aminobutyric Acid (GABA)/NAA levels will show a greater increase after 1 week, in uridine-treated vs. placebo-treated veterans with suicidal ideation.
  Proton-1 Magnetic Resonance Spectroscopy (1H-MRS) is a safe and non-invasive method for in-vivo measurement of brain chemistry relevant to mental health, including the neurotransmitters, glutamate, glutamine, and GABA.
Time Frame: 1 week
Population: Statistical outliers and motion-corrupted neuroimaging data were removed from this analysis.
Measure: Mean (Standard Deviation); unit: ratio of GABA/NAA
Arm/Group | Uridine | Placebo
Number analyzed (Participants) | 31 | 33
ratio of GABA/NAA | 0.00113 (0.0327) | 0.00564 (0.0279)

4. Secondary Outcome: Change From Baseline in Brain Total Choline/N-acetylaspartate (NAA) Levels, Measured With Proton-1 Magnetic Resonance Spectroscopy (1H-MRS) Neuroimaging
Description: Proton-1 Magnetic Resonance Spectroscopy (1H-MRS) is a safe and non-invasive method for in-vivo measurement of brain chemistry relevant to mental health, including the neurometabolites, choline and N-acetylaspartate.
Time Frame: 1 week
Population: Statistical outliers and motion-corrupted neuroimaging data were removed from this analysis.
Measure: Mean (Standard Deviation); unit: ratio of tCho/NAA
Arm/Group | Uridine | Placebo
Number analyzed (Participants) | 31 | 33
ratio of tCho/NAA | 0.00461 (0.012) | -0.00117 (0.0106)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Uridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/38
Other Adverse Events (participants affected / at risk) | 21/37 | 27/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uridine (N=37) | Placebo (N=38)
Suicidal Ideation/Behavior (Psychiatric disorders) | 0 | 1 — The participant completed treatment but missed the final visit. Staff learned they were hospitalized for suicidal ideation, opioid withdrawal, and methamphetamine-induced psychosis. Their history included 7 attempts, 2 interrupted, and 5 aborted.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Uridine (N=37) | Placebo (N=38)
Abdominal cramp, Nausea, Indigestion, Diarrhea (Gastrointestinal disorders) | 13 | 14
Headache, lightheadedness (Nervous system disorders) | 5 | 6
Psychiatric (Psychiatric disorders) | 2 | 4
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03265964/Prot_SAP_000.pdf